CLINICAL TRIAL: NCT00004368
Title: Phase I Study of Colchicine Therapy in Childhood Hepatic Cirrhosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Children's Hospital Colorado (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11947; CHD-1089
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Cirrhosis; Liver Cirrhosis
Keywords: hepatic cirrhosis; gastrointestinal disorders; rare disease
MeSH Terms: conditions — Fibrosis; Liver Cirrhosis; Gastrointestinal Diseases; Rare Diseases | interventions — Colchicine

INTERVENTIONS:
Drug: colchicine

SUMMARY:
OBJECTIVES:

I. Investigate the efficacy and safety of colchicine therapy in improving hepatic function and reducing hepatic fibrosis (scarring) in children with hepatic cirrhosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive colchicine orally twice daily for 24 months. After the first month, the dose of colchicine will increase and remain at that dose for the duration of study.

Patients are evaluated every 6 months during study.

ELIGIBILITY:
* Advanced hepatic fibrosis or cirrhosis in children
* Not pregnant

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15
Dates: Start 1990-05

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J. Sokol, Study Chair — Children's Hospital Colorado